CLINICAL TRIAL: NCT04148976
Title: Effect of Dietary Intervention on LDL-C Levels and Lipoprotein Subclasses Distribution in Patients With Hypercholesterolemia
Brief Title: Effect of Dietary Intervention on LDL-C and Lipoprotein Subclasses Distribution in Patients With Hypercholesterolemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Nimbe Torres y Torres, Nimbe Torres y Torres, PhD, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 706
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Hypercholesterolemia; Disease; Dyslipidemias
Keywords: hypercholesterolemia; dietary portfolio; soy protein; LDL-C; lipoprotein subclasses; nopal; chia seed; functional foods
MeSH Terms: conditions — Hypercholesterolemia; Disease; Dyslipidemias

STUDY DESIGN:
Intervention Model Description: This study had two stages. In the first stage, subjects underwent dietary standardization with low saturated fat dietary treatments (LSFD) designed according to NCEP, ATP III criteria, and that provided the same amount of energy as that of the habitual diet of the volunteers, as assessed by 24-hour dietary recalls.
  In the second stage, subjects were randomly allocated to two different treatments, 1) LSFD plus placebo or, 2) LSFD plus dietary portfolio. Subjects were instructed to consume two packets of the corresponding treatment a day dissolved in 250-300 ml of water before breakfast and dinner for two consecutive months.
Who Masked: Participant, Investigator
Masking Description: The DP and placebo were packed in identical form and appearance. The treatment was provided in sealed boxes to the participants by an individual external to the study, but who performed the randomization. Furthermore, the researcher and the volunteer were unaware of the allocation of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (P) (Placebo Comparator): The placebo consisted of 30g of calcium caseinate, 30g of maltodextrin, and 0.2g of flavoring. The placebo was provided in a dehydrated form in a packet containing 30g each provided twice a day. The content of each packet was dissolved in 250ml of water.
  Interventions: Dietary Supplement: Placebo
- Dietary Portfolio (DP) (Experimental): The DP included 25g of soy protein, 14g of dehydrated nopal,14g of oats, 4g of chia seeds, 4g of inulin, and 0.15g of flavoring. The DP was provided in a dehydrated form in a packet containing 30g each. The content of each packet was dissolved in 250ml of water.
  Interventions: Dietary Supplement: Dietary portfolio

INTERVENTIONS:
Dietary Supplement: Placebo — A mixture of maltodextrins and calcium caseinate divided into 30g individual packets.
  Arms: Placebo (P)
Dietary Supplement: Dietary portfolio — A mixture of functional foods divided into 30g individual packets.
  Arms: Dietary Portfolio (DP)

SUMMARY:
The primary aim of the present study was to elucidate the effect of a combination of functional foods on the low-density lipoprotein cholesterol (LDL-C) levels and on the distribution of the lipoprotein subclasses in subjects with hypercholesterolemia. To accomplish the latter, subjects that met the inclusion criteria and had mild hypercholesterolemia (Total cholesterol >200mg/dL, and LDL-C >130mg/dL <190 mg/dL) were recruited for double-blind, parallel, controlled dietary intervention study. After two weeks of dietary standardization with an isocaloric diet, subjects were randomized and allocated to either placebo or a dietary portfolio treatment for two months. The secondary endpoints were the size of the different lipoprotein subclasses, total cholesterol levels, high density -lipoprotein cholesterol (HDL-C) levels, apolipoprotein B, triglycerides, total/HDL-C ratio, apolipoprotein B/apolipoprotein A ratio, and anthropometric measurements.

DETAILED DESCRIPTION:
The present work took place at the Department of Physiology of Nutrition at the Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (INCMNSZ). The study followed a randomized, controlled, double-blind, parallel design encompassing five visits. On the first visit, volunteers were screened for eligibility criteria. Subjects that met the inclusion criteria were then invited to a second visit. Herein, volunteers received a thorough explanation of the experimental maneuver, as well as the overall objectives of the study. Thereafter, subjects who agreed to participate signed a consent form.

Upon agreement, assessment of habitual dietary intake and physical activity was obtained by 24-hour dietary recalls, food frequency questionnaire (FFQ), and by the International Physical Activity Questionnaire (IPAQ), respectively. Additionally, anthropometric measurements and blood samples were registered and collected. Then, volunteers underwent dietary standardization for two weeks with isocaloric diets (LSFD), which followed the National Cholesterol Education Program (NCEP) , Adult Treatment Panel III (ATP III) criteria. That is, 50-60% carbohydrates, 15% protein, 25-35% fat,<7% saturated fat,≤ 200mg of dietary cholesterol, 20-35g of fiber, and 2000mg/d of sodium.

On the third visit, subjects were randomly allocated to either LSFD plus placebo or an LSFD plus the dietary portfolio (DP). Of note, the prescribed diets were matched to the volunteers' habitual caloric intake -considering the energy provided by the placebo or DP- to avoid variability of the endpoint variables due to weight-loss. The DP and placebo provided 200kcal; the DP included 25g of soy protein, 14g of dehydrated nopal,14g of oats, 4g of chia seeds, 4g of inulin, and 0.15g of flavoring. The placebo consisted of 30g of calcium caseinate, 30g of maltodextrin, and 0.2g of flavoring. The organoleptic characteristics and packaging were similar between treatments. Subjects were instructed to consume two packets per day, preferably with breakfast and dinner. The content of each packet (30g of product) was dissolved in 250-300ml of water.

Volunteers followed the given treatment for two consecutive months, during which two follow-up visits took place. Blood samples, anthropometric characteristics, and blood pressure were obtained in all visits.

Compliance to diet, placebo, and DP was assessed with 24-hour dietary recalls, 3-day dietary records, and with the number of empty packets returned on the corresponding visits.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Body mass index (BMI) 25 to ≤ 39.9 kg/m2
* Adults between 20 and 60 years of age
* Total cholesterol levels of >200mg/dL in serum
* LDL-C levels ≥130mg/dL ≤190mg/dL
* Literate subjects
* Signature of informed consent

Exclusion Criteria:

* Subjects with diabetes
* Diseases that produce obesity or diabetes
* Cardiovascular events
* Weight-loss of ≥ 3kg on the preceding months to the study
* Catabolic diseases such as cancer and acquired immunodeficiency syndrome
* Pregnancy and breastfeeding
* Positive Smoking
* Pharmacological treatment including:

Antihypertensive drugs Hypoglycemic agents Statins, fibrates or any other treatment for dyslipidemia Steroid medications Chemotherapy, immunosuppressants, and radiotherapy Anorexigens or other medication to induce weight-loss

* Subjects with high cardiovascular risk
* Subjects with symptomatic digestive pathologies

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2013-02-28 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Low density lipoprotein- cholesterol (LDL-C) | Change in total LDL-C after 2.5 months of treatment
  Plasma total LDL-C (mg/dl)
Lipoprotein subclasses | Change in small, medium and large LDL, HDL and VLDL lipoprotein subclasses after 2.5 months of treatment
  High density lipoprotein (HDL), low density lipoprotein (LDL), and very low density lipoprotein (VLDL) subclasses (small medium and large) as measure by nuclear magnetic resonance spectroscopy (NMR) in μmol/L.

SECONDARY OUTCOMES:
Total cholesterol | Change in total cholesterol after 2.5 months of treatment
  Plasma total cholesterol (mg/dL)
Triglycerides | Change in triglycerides after 2.5 months of treatment
  Plasma triglycerides (mg/dL)
High density lipoprotein cholesterol (HDL-C) | Change after 2.5 months of treatment
  Plasma HDL cholesterol (mg/dL)
Apolipoprotein B | Change after 2.5 months of treatment
  Change in apolipoprotein B in
Apolipoprotein A | Change after 2.5 months of treatment
  Change in apolipoprotein A in plasma
Total/ high density lipoprotein cholesterol (HDL-C) ratio | Change after 2.5 months of treatment
  Change in total/ high density lipoprotein cholesterol (HDL-C) ratio
Apolipoprotein B/Apolipoprotein A ratio | Change after 2.5 months of treatment
  Change in Apolipoprotein B / Apolipoprotein A ratio

CONTACTS AND LOCATIONS:
Overall Officials: Nimbe Torres y Torres, PhD, Principal Investigator — INCMNSZ

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guevara-Cruz M, Tovar AR, Aguilar-Salinas CA, Medina-Vera I, Gil-Zenteno L, Hernandez-Viveros I, Lopez-Romero P, Ordaz-Nava G, Canizales-Quinteros S, Guillen Pineda LE, Torres N. A dietary pattern including nopal, chia seed, soy protein, and oat reduces serum triglycerides and glucose intolerance in patients with metabolic syndrome. J Nutr. 2012 Jan;142(1):64-9. doi: 10.3945/jn.111.147447. Epub 2011 Nov 16. PMID 22090467
- [Background] Guevara-Cruz M, Flores-Lopez AG, Aguilar-Lopez M, Sanchez-Tapia M, Medina-Vera I, Diaz D, Tovar AR, Torres N. Improvement of Lipoprotein Profile and Metabolic Endotoxemia by a Lifestyle Intervention That Modifies the Gut Microbiota in Subjects With Metabolic Syndrome. J Am Heart Assoc. 2019 Sep 3;8(17):e012401. doi: 10.1161/JAHA.119.012401. Epub 2019 Aug 27. PMID 31451009
- [Background] Jenkins DJ, Josse AR, Wong JM, Nguyen TH, Kendall CW. The portfolio diet for cardiovascular risk reduction. Curr Atheroscler Rep. 2007 Dec;9(6):501-7. doi: 10.1007/s11883-007-0067-7. PMID 18377791
- [Background] Mora S, Otvos JD, Rifai N, Rosenson RS, Buring JE, Ridker PM. Lipoprotein particle profiles by nuclear magnetic resonance compared with standard lipids and apolipoproteins in predicting incident cardiovascular disease in women. Circulation. 2009 Feb 24;119(7):931-9. doi: 10.1161/CIRCULATIONAHA.108.816181. Epub 2009 Feb 9. PMID 19204302
- [Background] Torres N, Guevara-Cruz M, Granados J, Vargas-Alarcon G, Gonzalez-Palacios B, Ramos-Barragan VE, Quiroz-Olguin G, Flores-Islas IM, Tovar AR. Reduction of serum lipids by soy protein and soluble fiber is not associated with the ABCG5/G8, apolipoprotein E, and apolipoprotein A1 polymorphisms in a group of hyperlipidemic Mexican subjects. Nutr Res. 2009 Oct;29(10):728-35. doi: 10.1016/j.nutres.2009.09.013. PMID 19917453
- [Background] Ascencio C, Torres N, Isoard-Acosta F, Gomez-Perez FJ, Hernandez-Pando R, Tovar AR. Soy protein affects serum insulin and hepatic SREBP-1 mRNA and reduces fatty liver in rats. J Nutr. 2004 Mar;134(3):522-9. doi: 10.1093/jn/134.3.522. PMID 14988441
- [Background] Lopez-Romero P, Pichardo-Ontiveros E, Avila-Nava A, Vazquez-Manjarrez N, Tovar AR, Pedraza-Chaverri J, Torres N. The effect of nopal (Opuntia ficus indica) on postprandial blood glucose, incretins, and antioxidant activity in Mexican patients with type 2 diabetes after consumption of two different composition breakfasts. J Acad Nutr Diet. 2014 Nov;114(11):1811-8. doi: 10.1016/j.jand.2014.06.352. Epub 2014 Aug 12. PMID 25132122
- [Background] Medina-Vera I, Sanchez-Tapia M, Noriega-Lopez L, Granados-Portillo O, Guevara-Cruz M, Flores-Lopez A, Avila-Nava A, Fernandez ML, Tovar AR, Torres N. A dietary intervention with functional foods reduces metabolic endotoxaemia and attenuates biochemical abnormalities by modifying faecal microbiota in people with type 2 diabetes. Diabetes Metab. 2019 Apr;45(2):122-131. doi: 10.1016/j.diabet.2018.09.004. Epub 2018 Sep 25. PMID 30266575
- [Derived] Vazquez-Manjarrez N, Guevara-Cruz M, Flores-Lopez A, Pichardo-Ontiveros E, Tovar AR, Torres N. Effect of a dietary intervention with functional foods on LDL-C concentrations and lipoprotein subclasses in overweight subjects with hypercholesterolemia: Results of a controlled trial. Clin Nutr. 2021 May;40(5):2527-2534. doi: 10.1016/j.clnu.2021.02.048. Epub 2021 Mar 6. PMID 33932799